CLINICAL TRIAL: NCT01051544
Title: Randomised Study of First TIME Immunotolerance Induction in Patients With Severe Type A Haemophilia With Inhibitor at High Risk of Failure: Comparison of Induction of Immune Tolerance With FVIII Concentrates With or Without Von Willebrand Factor Acronym: RES.I.S.T.- Naive
Brief Title: Study of First TIME Immunotolerance Induction in Severe Hemophilia A Patients With Inhibitor at High Risk of Failure: Comparison With FVIII Concentrates With or Without Von Willebrand Factor - RES.I.S.T. Naive
Acronym: RESIST NAIVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: complete per PI
Sponsor: City of Hope Medical Center (Other)
Collaborators: Charta Foundation (Other); Grifols Biologicals, LLC (Industry); CSL Behring (Industry); Biotest Pharmaceuticals Corporation (Industry); Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06201; 2008-007016-15 (EudraCT Number)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
Keywords: ITI; HAEMOPHILIA A; INHIBITORS; VWF/FVIII Concentrates
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; recombinant factor VIII SQ; optivate; factor VIII, von Willebrand factor drug combination; von Willebrand Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- von Willebrand factor-free FVIII concentrates (Active Comparator): Patients treated with FVIII concentrates
  Interventions: Drug: FVIII Concentrates
- FVIII/VWF concentrates (Active Comparator): Patients treated with FVIII/VWF concentrates
  Interventions: Drug: FVIII/VWF concentrates

INTERVENTIONS:
Drug: FVIII Concentrates — Patients will be centrally randomized to receive a von Willebrand factor-free FVIII concentrate (recombinant or plasma-derived, monoclonally-purified). The choice of product brand will be based on physician / patients preferences.
  Other Names: Including but not limited to:; Advate; Beriate P; Hemofil M; Helixate; Kogenate; Kogenate SF; Monarch M; Monoclate; Recombinate; Refacto; Replenate; Xyntha
  Arms: von Willebrand factor-free FVIII concentrates
Drug: FVIII/VWF concentrates — Patients will be centrally randomized to receive a FVIII/VWF concentrate of 200 IU/Kg by one or two bolus injections daily.The choice of product brand will be based on physician / patients preferences.
  Other Names: Including but not limited to:; Koate-DVI; 8Y; Optivate; Alphanate; Fahndi; Haemate P; Humate P; Haemoctine SDH; Octanate; Wilate; Emoclot DI; Factane
  Arms: FVIII/VWF concentrates

SUMMARY:
This is a prospective, controlled, randomized, open label study, aimed at comparing FVIII/VWF concentrates with FVIII concentrates at 200 IU/kg daily in their ability to induce immune tolerance in Haemophilia A patients with high responding inhibitors and poor prognosis for success.

DETAILED DESCRIPTION:
The presence of Factor VIII (FVIII) inhibitor prevents FVIII infusions from working properly and makes treatment of bleeding episodes very difficult. Having an inhibitor is a serious and life-threatening complication in patients with Hemophilia. The usual treatment of patients with FVIII inhibitors involves "immune tolerance induction" (ITI). Immune Tolerance means that the body can accept infused FVIII and that FVIII is again effective in controlling bleeds. ITI involves giving high doses of FVIII regularly until the inhibitor disappears. This treatment is not always effective. The inhibitor persists in about 1 in 5 patients who undergo ITI.

There are 2 types of FVIII concentrates: FVIII concentrates derived from human plasma, which contain the von Willebrand factor, and concentrates of FVIII without VWF (recombinant or plasma derived). Both types of concentrates are commonly used to induce immune tolerance in patients with Hemophilia A. Retrospective studies in subjects with hemophilia and inhibitors at risk for failing ITI, have indicated a higher rate of success if patients were treated with von Willebrand containing factor VIII concentrates. It is not known whether the addition of Von Willebrand factor offers an advantage to achieving immune tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. severe hemophilia A (FVIII<1%);
2. male, any age;
3. high responders (peak inhibitor levels > 5 BU);
4. any inhibitor level at study enrolment;
5. ability and willingness to participate in the study;
6. at least one of the following risk factors for ITI failure:

   * peak inhibitor titer > 200 BU
   * titer at ITI start > 10 BU
   * age > 7 years
   * time between inhibitor occurrence and ITI > 2 years
7. absence of high risk of cardiovascular, cerebrovascular or other thromboembolic events as deemed by the treating clinician.

Exclusion Criteria:

1. concomitant systemic treatment with immunosuppressive drugs;
2. concomitant experimental treatment;
3. previous ITI attempt;
4. previous history of myocardial infarction and/or cerebral stroke.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Primary end point is the success in inducing immune tolerance, defined as: the abolition of the inhibitor to < 0.6 BU within 33 months of ITI with a factor VIII recovery ≥ 66% and half-life ≥ 6 hrs, and measured after a 72-hour washout period. | 33 months

SECONDARY OUTCOMES:
Absence of relapse, up to 12 months after achievement of Immune Tolerance | 12 months
Time to achieve partial or complete success as defined in the protocol. | 33 months
Safety Compliance to treatment | 33 months
Cost of Care | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia P Ewing, MD, Principal Investigator — Clinical Professor of Pediatrics, City of Hope National Medical Center, Dept. of Pediatrics, 1500 E. Duarte Rd. Duarte, CA 91010

REFERENCES:
- [Background] Berntorp E, Ekman M, Gunnarsson M, Nilsson IM. Variation in factor VIII inhibitor reactivity with different commercial factor VIII preparations. Haemophilia. 1996 Apr;2(2):95-9. doi: 10.1111/j.1365-2516.1996.tb00022.x. PMID 27214015
- [Background] Kreutz W: Immune tolerance induction (ITI) in Haemophilia A-patients with inhibitors - the choice of concentrate affecting success. Haematologica2001; 86 (S4):16-20
- [Background] Gringeri A, Musso R, Mazzucconi MG, Piseddu G, Schiavoni M, Pignoloni P, Mannucci PM; RITS-FITNHES Study Group. Immune tolerance induction with a high purity von Willebrand factor/VIII complex concentrate in haemophilia A patients with inhibitors at high risk of a poor response. Haemophilia. 2007 Jul;13(4):373-9. doi: 10.1111/j.1365-2516.2007.01484.x. PMID 17610550
- See also: Related Info — http://www.isth.org
- See also: Related Info — http://www.wfh.org
- See also: Related Info — http://www.eahad.org
- See also: Related Info — http://www.hemophilia.org
- See also: Related Info — http://www.aiceonline.it
- See also: Related Info — http://hematology.org
- See also: Related Info — http://www.aspho.org